CLINICAL TRIAL: NCT06657079
Title: A Combination of an Inhaled Budesonide and Ipratropium in Patients at Risk of Developing Acute Respiratory Distress Syndrome (ARDS): A Randomized Controlled Trial
Brief Title: A Combination of an Inhaled Budesonide and Ipratropium in Patients at Risk of Developing ARDS
Acronym: BUDIPRA-ARDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Badr University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Budesonide-Ipratropium ARDS; Damanhour University (Other: Faculty of pharmacy)
Record Dates: First submitted 2024-10-19; First posted 2024-10-24 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: ARDS; Prevention and Control
Keywords: ARDS; Inhaled Budesonide; Inhaled Ipratropium
MeSH Terms: interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combined standard aerosolized doses of budesonide (0.5 mg/2 mL) and ipratropium bromide (500/2 mL) (Active Comparator): combined standard aerosolized doses of budesonide (0.5 mg/2 mL) every 12 hours and ipratropium bromide (500/2 mL) every eight hours for up to five days
  Interventions: Drug: combined standard aerosolized doses of budesonide (0.5 mg/2 mL) every 12 hours and ipratropium bromide (500/2 mL) every eight hours for up to five days
- placebo (4 mL normal saline) (Placebo Comparator): placebo (4 mL normal saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: combined standard aerosolized doses of budesonide (0.5 mg/2 mL) every 12 hours and ipratropium bromide (500/2 mL) every eight hours for up to five days — combined standard aerosolized doses of budesonide (0.5 mg/2 mL) every 12 hours and ipratropium bromide (500/2 mL) every eight hours for up to five days
  Arms: combined standard aerosolized doses of budesonide (0.5 mg/2 mL) and ipratropium bromide (500/2 mL)
Drug: Placebo — Saline inhaler
  Arms: placebo (4 mL normal saline)

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a severe lung condition with high morbidity and mortality, despite advances in medical care. It involves an intense inflammatory response in the lungs, leading to endothelial damage, increased capillary permeability, and fluid accumulation, causing hypoxemia and respiratory failure. ARDS can result from various pulmonary and non-pulmonary triggers.

The 2012 Berlin criteria are widely used to diagnose ARDS, based on clinical signs, blood gas analysis, and chest imaging. The Lung Injury Prediction Score (LIPS) is used in emergency departments to assess the risk of ARDS, with scores of 4 or higher indicating a significant risk. Oxygenation impairment, particularly measured by the S/F ratio (oxygen saturation to inspired oxygen), is a strong predictor of ARDS. Common causes of death include severe hypoxemia, sepsis, organ failure, and respiratory complications.

ARDS treatment emphasizes supportive care, including lung-protective ventilation, prone positioning, and conservative fluid management. Pharmacological approaches have shown mixed results, with treatments like statins, surfactants, anticoagulants, and β2-agonists (e.g., salbutamol) offering inconsistent benefits.

Corticosteroids have demonstrated improvements in oxygenation in conditions that progress to ARDS. Inhaled corticosteroids are being explored to minimize systemic side effects by targeting the lungs directly. Ipratropium bromide, an inhaled bronchodilator, may also offer therapeutic benefits by reducing lung inflammation and pulmonary edema. However, it carries risks such as dry mouth, blurred vision, and potential cardiovascular side effects.

This double-blinded randomized controlled trial examines the effectiveness of early inhaled corticosteroids and ipratropium in reducing the risk of acute respiratory distress syndrome (ARDS) and its complications in high-risk patients. Participants will be administered aerosolized budesonide and ipratropium or a placebo every eight hours for five days. The primary outcome is the change in the oxygen saturation to inspired oxygen fraction ratio (S/F) after five days, assessing pulmonary oxygenation. Secondary outcomes include the incidence of ARDS, need for mechanical ventilation, length of hospital stay, and mortality. The study aims to evaluate whether early inhaled therapy can effectively prevent or alleviate ARDS, given the limited availability of pharmacological treatments for the condition.

DETAILED DESCRIPTION:
ARDS is a severe form of lung injury that continues to present high morbidity and mortality rates despite progress in diagnostic and therapeutic approaches. It is characterized by an intense inflammatory response in the lungs, leading to damage to the pulmonary endothelial and epithelial layers, increased permeability, and the development of pulmonary edema. These changes result in severe hypoxemia and acute respiratory failure. ARDS can be triggered by various factors, including pulmonary and non-pulmonary injuries.

Diagnosing ARDS is challenging due to the lack of a single definitive test. The Berlin criteria, which encompass clinical presentation, arterial blood gas analysis (PF ratio), and chest imaging, are widely utilized. The Lung Injury Prediction Score (LIPS) assists in evaluating ARDS risk, with a score of 4 or higher indicating increased likelihood.

Major causes of mortality in ARDS include persistent hypoxemia, sepsis, multiple organ failure, and respiratory failure. The management of ARDS primarily focuses on supportive care with the goal of mitigating lung injury by addressing underlying causes. Key strategies include employing lung-protective ventilation, prone positioning, and conservative fluid management. Pharmacologic treatments for ARDS have generally been unsuccessful in improving survival rates. Trials of therapies such as statins, aspirin, and vitamin D supplementation have not shown significant improvements in ARDS outcomes. β2-agonists have been investigated for their potential to enhance alveolar fluid clearance, but results have been inconsistent.

Corticosteroids have shown potential in improving oxygenation and histologic lung injury in ARDS. To maximize benefits while minimizing risks, corticosteroids should be administered within the first 14 days of ARDS diagnosis. Inhaled corticosteroids and ipratropium bromide are being explored as treatments for ARDS due to their targeted action on the respiratory system and reduced systemic side effects. Inhaled budesonide has shown potential in improving lung function and cytokine profiles. Ipratropium bromide, a short-acting anticholinergic bronchodilator, helps relax smooth muscles in the respiratory tract and is used in mechanically ventilated patients.

This study aims to assess the efficacy of inhaled corticosteroids and ipratropium bromide, in combination with standard care, in improving oxygenation, reducing ARDS incidence, minimizing the need for mechanical ventilation, shortening hospital stays, and lowering mortality rates. The potential benefits of these therapies in the prevention and management of ARDS are under investigation.

This study was structured as a double-blind, randomized clinical trial. It will be conducted in the ICU of a governmental hospital. Eligible participants are adults aged 18 years or older admitted through the emergency department. All participants will have least one risk factor for ARDS, a Lung Injury Prediction Score (LIPS) of 4 or more. Exclusion criteria includes pregnant patients, those unable to provide consent within 12 hours of hospital admission, or individuals with contraindications to corticosteroids or ipratropium, patients who had used inhaled corticosteroids or muscarinic antagonists within the past 7 days, had ARDS onset prior to enrollment, or required mechanical ventilation before admission. Those with an expected hospital stay of less than 48 hours, poor prognosis, or admitted for palliative care will not be included in the trial. Participants will be randomized in a 1:1 ratio within 12 hours of presentation. This trial was approved by the BUC-Institutional Ethical Committee (No. BUC-IACUC-240318-80). All patients agree to participation will sign a participation consent.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)

  * Admitted through the ED with at least one known risk factor for ARDS
  * A LIPS greater than or equal to 4, and acute hypoxemia (defined as at least 2 L/min of supplemental oxygen requirement to maintain an oxygen saturation between 92% and 98%).

Exclusion Criteria:

* Pregnant patients

  * Inability to obtain consent within 12 hours of hospital presentation
  * Indications or contraindications for either corticosteroids or ipratropium (allergy to either budesonide and/or ipratropium bromide use
* History of asthma or chronic obstructive lung disease

  * ECG and/or clinical presentation suggestive of acute coronary ischemia
  * A new cardiac arrhythmia including atrial fibrillation
  * Uncontrolled atrial fibrillation; or persistent sinus tachycardia of >130/minute
  * Receipt of inhaled muscarinic antagonist or corticosteroids in prior 7 days
  * Systemic steroid treatment on admission or within 7 days prior to admission equivalent to more than 5 mg of prednisone daily
  * Onset of ARDS (by Berlin criteria including noninvasive ventilation) prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was longitudinal change in the S/F | change in the S/F for up to 5 days

SECONDARY OUTCOMES:
progression to ARDS | Through the ICU stay up to 28 day
  Final diagnosis of ARDS was determined using Berlin criteria after chest radiograph.
  5. Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R,

CONTACTS AND LOCATIONS:
Overall Officials: amira B kassem, Principal Investigator — Damanhour University
Locations (1):
- Mashtoul El Souq governmental hospital (50 beds), Sharkia, Egypt, Cairo, Egypt